CLINICAL TRIAL: NCT01794676
Title: A Pilot Study of Genetic Evaluation of Families With Endocrine Cancers
Brief Title: Genetic Evaluation of Families With Endocrine Cancers
Acronym: MEN1
Status: Completed | Type: Observational
Sponsor: Jersey Shore University Medical Center (Other)
Collaborators: Rutgers University (Other); Rutgers Cancer Institute of New Jersey (Other)
Responsible Party: Principal Investigator, Alexander Shifrin, MD, FACS, FACE, Attending Endocrine Surgeon, Jersey Shore University Medical Center
Other Study IDs: IIU03-07; MEN1 (Other: Jersey Shore University Medical Center)
Record Dates: First submitted 2013-02-15; First posted 2013-02-20 (Estimated); Last update posted 2017-06-16 (Actual); Status verified 2017-06

CONDITIONS: Pancreatic Cancer; Thymic Cancer; Parathyroid Disease; MEN1 Syndrome
Keywords: Pancreatic cancer; Thymic cancer; Parathyroid disease; MEN1 syndrome; Genomic DNA; MEN1 gene sequence
MeSH Terms: conditions — Pancreatic Neoplasms; Thymus Neoplasms; Parathyroid Diseases; Multiple Endocrine Neoplasia Type 1 | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Approximately 10 ml of blood will be drawn from each participant. Tumor samples will be obtained from any prior surgeries, if available.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Family 1: Approximately a 10 ml of blood draw will be taken from each participant for genetic testing.
  Interventions: Genetic: Blood draw
- Family 2: Approximately a 10 ml of blood draw will be taken from each participant for genetic testing.
  Interventions: Genetic: Blood draw
- Family 3: Approximately a 10 ml of blood draw will be taken from each participant for genetic testing.
  Interventions: Genetic: Blood draw

INTERVENTIONS:
Genetic: Blood draw — Blood draw

SUMMARY:
This study is being conducted to identify altered genetic factors that may exist and influence endocrine cancers in unrelated MEN1 families with different cancers. A grading system will be developed for endocrine cancers, including pancreatic cancers, thymus gland cancers, parathyroid disease and MEN1 syndrome as low-risk and high-risk to improve screening and timing of surgery.

DETAILED DESCRIPTION:
Participants will be sent a personal medical questionnaire and family history questionnaire to complete prior to their visit. Participants will meet with a genetic counselor face-to-face for up to 120 minutes to complete a personal and family history. Participants will receive genetic counseling including education about MEN1 syndrome and recommendations for the management of this disease. The genetic counselor will also assist participants with coping mentally. The genetic counselor will review the risk, benefits and limitations of genetic testing.

After study eligibility is confirmed and the participant agrees to participate in the study, approximately 10 ml (2 teaspoons) of blood will be taken from the participant for genetic testing. Tumor samples from any prior surgeries will be requested from the Jersey Shore University Medical Center pathology department for review.

The participant's blood sample and any tumor samples will be assigned a unique identifier. Participants will not be identified by name. This identifier, along with the participant's age, sex, ethnicity and if applicable, age of cancer diagnosis (or MEN1 syndrome diagnosis) will be kept at Jersey Shore University Medical Center research department. Medical records will be reviewed for demographics, known cancer risk factors, family history, age and stage at diagnosis of disease, tumor characteristics, previous and current treatments, medication history, test and study results, and pathology/surgery reports. Blood and tumor samples will be sent to the Functional Genomics Facility at The Cancer Institute of New Jersey and Rutgers University Cell & DNA Repository for processing and/or analysis to identify the genetic pattern in patients at risk for MEN1.

The result of the genetic test for the MEN1 gene will be provided to the participant by either the genetic counselor or study doctor. The genetic counselor or study doctor will interrupt the results for the participant and provide emotional support, if necessary. The results of any altered genes will not be disclosed to the participant.

Medical records will be reviewed annually to determine the status of the participant's disease, if any. Participants will be contacted directly by phone or in person at follow-up clinic visit(s) for the collection of information not recorded in the participant's medical record for up to 20 years.

ELIGIBILITY:
Eligibility Criteria:

* Age ≥ 13 years.
* A signed written informed consent
* Existing patients and their family members of Investigators with MEN1 syndrome.
* Willing to undergo venipuncture to obtain 10 ml of blood and complete genetic counseling and informed consent process.

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Individuals belonging to families observed with MEN1 mutation related cancers.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2013-03; Primary Completion 2015-09 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Modified genetic factors that exist and may influence the phenotypic presentation of disease in unrelated MEN 1 families. | Within 3 Months from blood draw
  To identify modifying genetic factors that exist and that may influence phenotypic presentation of the disease in unrelated MEN 1 families with different clinical presentation of the disease.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Shifrin, MD, Principal Investigator — Jersey Shore University Medical Center
Locations (1):
- Jersey Shore University Medical Center, Neptune City, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1) Multiple Endocrine Neoplasia Type 1 (MEN1) Syndrome. Marini F, Falchetti A, Luzi E, Tonelli F, Maria Luisa B. In: Riegert-Johnson DL, Boardman LA, Hefferon T, Roberts M, editors. Cancer Syndromes [Internet]. Bethesda (MD): National Center for Biotechnology Information (US); 2009-.2008 Jul 18 2) Multiple endocrine neoplasia. White ML, Doherty GM. Surg Oncol Clin N Am. 2008 Apr;17(2):439-59 3) Multiple endocrine neoplasia type 1 (MEN1). Thakker RV. Best Pract Res Clin Endocrinol Metab. 2010 Jun; 4) Guidelines for diagnosis and therapy of MEN type 1 and type 2. Brandi ML, Gagel RF, Angeli A, Bilezikian JP, Beck-Peccoz P, Bordi C, Conte-Devolx B, Falchetti A, Gheri RG, Libroia A, Lips CJ, Lombardi G, Mannelli M, Pacini F, Ponder BA, Raue F, Skogseid B, Tamburrano G, Thakker RV, Thompson NW, Tomassetti P, Tonelli F, Wells SA Jr, Marx SJ. J Clin Endocrinol Metab. 2001 Dec;86(12):5658-71. 5) Multiple endocrine neoplasia type 1 (MEN1) germline mutations in familial isolated primary hyperparathyroidism. Pannett AA, Kennedy AM, Turner JJ, Forbes SA, Cavaco BM, Bassett JH, Cianferotti L, Harding B, Shine B, Flinter F, Maidment CG, Trembath R, Thakker RV. Clin Endocrinol (Oxf). 2003 May;58(5):639-46. 6) Human Gene Mutation Database, http://www.hgmd.org/ 6) Human Gene Mutation Database, http://www.hgmd.org/ 7) Familial isolated primary hyperparathyroidism caused by mutations of the MEN1 gene. Hannan FM, Nesbit MA, Christie PT, Fratter C, Dudley NE, Sadler GP, Thakker RV. Nat Clin Pract Endocrinol Metab. 2008 Jan; 8) Familial isolated hyperparathyroidism: clinical and genetic characteristics of 36 kindreds. Simonds WF, James-Newton LA, Agarwal SK, Yang B, Skarulis MC, Hendy GN, Marx SJ. Medicine (Baltimore). 2002 Jan;81(1):1-26. 9) Genotype-phenotype analysis in multiple endocrine neoplasia type 1. Kouvaraki MA, Lee JE, Shapiro SE, Gagel RF, Sherman SI, Sellin RV, Cote GJ, Evans DB. Arch Surg. 2002 Jun;137(6):641-7.